CLINICAL TRIAL: NCT06784310
Title: Feeding the Family: Nutrition Security Intervention to Improve Physical and Mental Health Among Low-resource Families
Brief Title: Food Insecurity, Social Determinants of Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alison Gustafson (Other)
Responsible Party: Sponsor-Investigator, Alison Gustafson, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 96706
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Food Insecurity; Type 2 Diabetes Mellitus (T2DM); Hypertension
Keywords: Food as medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A randomized trial with a 2x2 design and a delayed control comparison group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MTM (medically tailored meals) (Active Comparator): Fully prepared meals are delivered on a weekly basis, and tailored to specific health needs
  Interventions: Behavioral: Medically Tailored Meals; Behavioral: Nutritional Counseling
- GP (grocery prescription) (Active Comparator): cards are issued to each participant per month to be spent on eligible healthy food items
  Interventions: Behavioral: Grocery Prescription; Behavioral: Nutritional Counseling
- MTM + GP (medically tailored meals and grocery prescription) (Active Comparator): delivered weekly MTM meals and the GP monthly grocery funds
  Interventions: Behavioral: Medically Tailored Meals and Grocery Prescription; Behavioral: Nutritional Counseling
- Nutrition Counseling (Placebo Comparator): 30 minutes per week of nutrition counseling and assistance. This group will receive the Grocery Prescription package after the last set of study measures are completed
  Interventions: Behavioral: Nutritional Counseling

INTERVENTIONS:
Behavioral: Medically Tailored Meals — Dare to Care will provide meals each week for 12 weeks tailored for comorbidities. Meals will be provided to both the adult and the child(ren). Meals have been developed with a Registered Dietitian and have been approved through Food Is Medicine Coalition (FMIC). Meals are delivered via Door Dash each week.
  Arms: MTM (medically tailored meals)
Behavioral: Grocery Prescription — Instacart Fresh Funds (for those that need delivery) or Kroger Grocery Rx cards will be issued to each participant per month to be spent on eligible healthy food items (lean protein, lean dairy, fruits, vegetables, eggs, and nuts). For each participating child in the household, they will receive additional funds/per child loaded on their grocery Rx card
  Arms: GP (grocery prescription)
Behavioral: Medically Tailored Meals and Grocery Prescription — will receive both tailored MTM meals per week for adult and child(ren) and the GP monthly grocery funds
  Arms: MTM + GP (medically tailored meals and grocery prescription)
Behavioral: Nutritional Counseling — 30 minutes per week of nutrition counseling and assistance.

SUMMARY:
Food is Medicine for the whole will test an intervention which provides medically tailored meals, or grocery voucher cards, or a combination of these food and nutrition resources to a caregiver and children living in the household. The study will examine how providing healthy tailored food and nutrition services can improve health outcomes, such as blood pressure and cholesterol levels.

DETAILED DESCRIPTION:
The proposal addresses the key goals of Humana Foundation related to, "Effective and equitable interventions to increase access to healthy diets promoting physical & mental health benefits". The interdisciplinary team comprised of clinicians, researchers in public health, nutrition, mental health, and community partners will evaluate the effectiveness of a whole family nutrition security intervention to provide evidence supporting key policies on reimbursement of health-related social needs (HRSN) as a medically covered benefit. The study team will use a user-centered approach to examine how to engage the whole family in the short-term, while creating a sustainable model for clinic and community partnerships to use in the long-term. This proposal aims to answer the question "How can a food as medicine choice model with tailored dose improve health outcomes across the family?". To answer this question, investigators are proposing a pragmatic randomized control trial (pRCT) using a 2X2 factorial design among Medicaid families, adults with children ages 5-18, with an adult diagnosed with either hypertension or Type 2 Diabetes (T2DM), child has a BMI categorized as obese or overweight, and report being food insecure. The pRCT will take place in Louisville, Kentucky with University of Louisville Health as the clinic provider, in an urban setting with a high percentage of adults reporting race/ethnicity as Black or African American. The community partners are Dare to Care Food Bank as the medically tailored meal (MTM) provider, and Kroger Health/Soda Health as the grocery prescription provider (GP).

ELIGIBILITY:
Inclusion Criteria:

* Have at least one child ages 6-17, inclusive, living in the household with the adult at least 50% of the time
* Diagnosis of stage 3 or 4 Hypertension in last 12 months, or diagnosis of T2DM in the last 12 months
* Experiencing food insecurity as indicated by 2-item Hunger Vital Sign
* English speaking
* No plans to move from the area for at least 1 year
* Willing and able to accept text messages
* Free living to the extent that participant has control over dietary intake
* Willing and able to provide written informed consent and participate in all study activities.

Exclusion Criteria:

* Participant in diabetes, nutrition, or weight research intervention in last 12 months
* Considering bariatric surgery in the next year or prior bariatric surgery
* Lack of safe, stable residence and ability to store meals
* Lack of telephone which can receive text messages
* Pregnancy/breastfeeding or intended pregnancy in the next year
* History of malignancy, other than non-melanoma skin cancer, unless surgically or medically cured > 5 years ago or in remission
* Advanced kidney disease (estimated creatinine clearance < 30 mL/min)
* Known drug or alcohol misuse in the past 2 years
* Known psychosis or major psychiatric illness that prevents participation with study activities
* Intermittent use of medications (e.g., oral or intravenous glucocorticoids) that are likely to affect blood sugar.

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) percentile - child | Baseline, post intervention (week 12), and month 6
  BMI percentile is automatically calculated in the Electronic Health Record (EHR) from height and weight using age- and gender-specific CDC growth charts
Change in body mass index percentile - adult | Baseline, post intervention (week 12), and month 6
  BMI percentile is automatically calculated in the Electronic Health Record from height and weight
Change in systolic blood pressure - child | Baseline, post intervention (week 12), and month 6
  blood pressure measurements will be taken from the electronic health record
Change in diastolic blood pressure - child | Baseline, post intervention (week 12), and month 6
  blood pressure measurements will be taken from the electronic health record
Change in systolic blood pressure - adult | Baseline, post intervention (week 12), and month 6
  blood pressure measurements will be taken from the electronic health record
Change in diastolic blood pressure - adult | Baseline, post intervention (week 12), and month 6
  blood pressure measurements will be taken from the electronic health record
Change in Hemoglobin A1c - child | Baseline, post intervention (week 12), and month 6
  A1c measures are collected at the clinic or affiliated lab and entered into the patient's EHR
Change in Hemoglobin A1c - adult | Baseline, post intervention (week 12), and month 6
  A1c measures are collected at the clinic or affiliated lab and entered into the patient's EHR
Change in total cholesterol - child | Baseline, post intervention (week 12), and month 6
  data will be pulled from the EHR
Change in total cholesterol - adult | Baseline, post intervention (week 12), and month 6
  data will be pulled from the EHR
Change in high-density lipoprotein (HDL) - child | Baseline, post intervention (week 12), and month 6
  data will be pulled from the EHR
Change in high-density lipoprotein (HDL) - adult | Baseline, post intervention (week 12), and month 6
  data will be pulled from the EHR
Change in low-density lipoprotein (LDL) - child | Baseline, post intervention (week 12), and month 6
  data will be pulled from the EHR
Change in low-density lipoprotein (LDL) - adult | Baseline, post intervention (week 12), and month 6
  data will be pulled from the EHR

SECONDARY OUTCOMES:
Change in Dietary Intake | Baseline, post intervention (week 12), and month 6
  Dietary intake is captured with the Dietary Screener Questionnaire (DSQ-10). Responses to these dietary intake questions are converted to daily cup equivalent estimates (e.g., 1.2 cups of vegetables per day, 1.1 cups of fruit per day, 2.3 cups of FVs per day) of daily FV intake. The 2020-2025 United States Dietary Guidelines for Americans recommend consuming 2 to 3 cups of vegetables per day and 1.5 to 2 cups of fruit per day.
Change in Family Stress | Baseline, post intervention (week 12), and month 6
  Anxiety and depression are measured using the Patient Health Questionnaire-4 (PHQ-4), a widely used and validated instrument. The PHQ-4 consists of a 2-question anxiety subscale and a 2-question depression subscale. For the anxiety subscale, respondents indicate how often, during the last 2 weeks, they have been bothered by the following: (1) feeling nervous, anxious, or on edge and (2) not being able to stop or control worrying. For the depression subscale, respondents indicate how often they have been bothered by the following: (1) little interest or pleasure in doing things and (2) feeling down, depressed, or hopeless. Response options for all four questions are as follows: not at all (0), several days (1), more than half the days (2), and nearly every day (3). For each of the subscales, zero is the minimum and a score of
  ‡ 3 is considered positive for screening purposes
Change in Nutrition Security | Baseline, post intervention (week 12), and month 6
  The one item Gretchen Swanson Nutrition Security question will be asked as follows:In the past month, how often did the participant worry that the food bought wouldn't provide enough nutrients for the family, even if the participant had enough to eat? Response options are never, rarely, sometimes, often, always, don't know
Change in Food Security | Baseline, post intervention (week 12), and month 6
  USDA 6-item food insecurity survey which can be found at this link https://www.ers.usda.gov/topics/food-nutrition-assistance/food-security-in-the-us/survey-tools Scores range from 0-6 with higher scores equating to lower food security

CONTACTS AND LOCATIONS:
Overall Officials: Alison Gustafson, PhD, MPH, RD, Principal Investigator — University of Kentucky
Locations (1):
- UofL Health, Louisville, Kentucky, United States